CLINICAL TRIAL: NCT01235546
Title: Cesarean Section Optimal Antibiotic Prophylaxis Trial
Brief Title: Study of Effectiveness and Safety of Azithromycin-based Extended-spectrum Prophylaxis to Prevent Post Cesarean Infection
Acronym: C/SOAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alan Tita (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Texas (Other); University of North Carolina (Other); Mission Hospital (Unknown); Ochsner Health System (Other); The University of Texas Health Science Center, Houston (Other); Columbia University (Other); University of Utah (Other); University of Mississippi Medical Center (Other)
Responsible Party: Sponsor-Investigator, Alan Tita, Professor, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: F090323006; NIH 1R01HD064729-01A1 (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Endometritis; Wound Infection; Abscess; Surgical Site Infection
Keywords: Pregnancy; Cesarean section; Antibiotic; Infections
MeSH Terms: conditions — Endometritis; Wound Infection; Abscess; Surgical Wound Infection; Infections | interventions — Azithromycin; Standard of Care; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo and standard of care (Placebo Comparator): 250 cc normal saline
  Interventions: Drug: Placebo and standard of care
- Azithromycin and Standard of care (Experimental): 500 mg Azithromycin in 250 cc normal saline
  Interventions: Drug: Azithromycin and standard of care

INTERVENTIONS:
Drug: Azithromycin and standard of care — 500 mg in 250 cc normal saline 1 time dose plus standard of care (cephazolin or clindamycin)
  Other Names: Zithromax
  Arms: Azithromycin and Standard of care
Drug: Placebo and standard of care — 250 cc normal saline, plus standard of care (cephazolin or clindamycin)
  Other Names: normal saline
  Arms: Placebo and standard of care

SUMMARY:
The Cesarean Section Optimal Antibiotic Prophylaxis (C/SOAP) study is a large pragmatic multi-center randomized clinical trial designed to evaluate the comparative effectiveness and safety of azithromycin-based extended-spectrum antibiotic prophylaxis (azithromycin plus standard narrow-spectrum cephalosporin) relative to standard single-agent cephalosporin (preferably prior to surgical incision) to prevent post-cesarean infection.

Hypothesis: Compared to narrow-spectrum prophylaxis (i.e. cefazolin alone, or clindamycin if cephalosporin allergy) prior to surgical incision, the addition of extended-spectrum prophylaxis (azithromycin + cefazolin) reduces the incidence of post-cesarean infection.

ELIGIBILITY:
Inclusion Criteria:

-

Pregnant Women aged 14 years and over at ≥ 24 weeks' viable gestation who will undergo unscheduled/non-elective cesareans with either:

1. Labor (spontaneous or induced): active labor (ongoing contractions and at least 4cm dilated or contractions for at least 4 hours with documented cervical change of ≥1cm dilatation or ≥50% effacement), or
2. Membrane rupture (standardized to duration of at least 4 hours prior to randomization).

Exclusion Criteria:

* Patient unwilling or unable to provide consent
* Multiple pregnancy
* Known azithromycin (or other macrolide) allergy
* Vaginal delivery
* Elective or scheduled cesarean prior to labor or membrane rupture.
* Azithromycin, erythromycin or other macrolide antibiotic use within 7 days of enrollment.
* Clinical chorioamnionitis or any other active bacterial infection (e.g. pyelonephritis, pneumonia, abscess) at time of randomization.
* Patient is unable or unlikely to follow-up after delivery (e.g. no prenatal care or a non-resident patient)
* Fetal demise or major congenital anomaly
* Significant liver disease defined as known cirrhosis or elevated transaminases of at least 3-fold upper limit of normal
* Significant renal disease defined as serum creatinine known to be >2.0 mg/dl or on dialysis.
* Active congestive heart failure (EF<45%) or pulmonary edema
* Active diarrhea at time of delivery
* Any patient with significant electrolyte abnormalities such as hypokalemia or hypocalcemia
* Any patient with structural heart disease or arrhythmias, or taking any medications known to prolong the QT interval
* Patient currently being treated with efavirenz, nelfinavir or fluconazole

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2013 (Actual)
Dates: Start 2011-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan TN Tita, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia University, New York, New York
  - Mission Hospital, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tita ATN, Rouse DJ, Blackwell S, Saade GR, Spong CY, Andrews WW. Emerging concepts in antibiotic prophylaxis for cesarean delivery: a systematic review. Obstet Gynecol. 2009 Mar;113(3):675-682. doi: 10.1097/AOG.0b013e318197c3b6. PMID 19300334
- [Background] Andrews WW, Hauth JC, Cliver SP, Savage K, Goldenberg RL. Randomized clinical trial of extended spectrum antibiotic prophylaxis with coverage for Ureaplasma urealyticum to reduce post-cesarean delivery endometritis. Obstet Gynecol. 2003 Jun;101(6):1183-9. doi: 10.1016/s0029-7844(03)00016-4. PMID 12798523
- [Background] Tita AT, Hauth JC, Grimes A, Owen J, Stamm AM, Andrews WW. Decreasing incidence of postcesarean endometritis with extended-spectrum antibiotic prophylaxis. Obstet Gynecol. 2008 Jan;111(1):51-6. doi: 10.1097/01.AOG.0000295868.43851.39. PMID 18165392
- [Derived] Martin JK, Longo SA, Jauk VR, Clark EAS, Saade GR, Boggess KA, Esplin S, Wapner RJ, Owens MY, Blackwell SC, Andrews WW, Szychowski JM, Tita AT. Neonatal outcomes in term and preterm infants following adjunctive azithromycin antibiotic prophylaxis for non-elective cesarean delivery. J Matern Fetal Neonatal Med. 2024 Dec;37(1):2367082. doi: 10.1080/14767058.2024.2367082. Epub 2024 Jun 14. PMID 38873885
- [Derived] Sanusi A, Ye Y, Boggess K, Saade G, Longo S, Clark E, Esplin S, Cleary K, Wapner R, Owens M, Blackwell S, Szychowski JM, Tita ATN, Subramaniam A. Timing of Adjunctive Azithromycin for Unscheduled Cesarean Delivery and Postdelivery Infection. Obstet Gynecol. 2022 Jun 1;139(6):1043-1049. doi: 10.1097/AOG.0000000000004788. Epub 2022 May 2. PMID 35675601
- [Derived] Boggess KA, Tita A, Jauk V, Saade G, Longo S, Clark EAS, Esplin S, Cleary K, Wapner R, Letson K, Owens M, Blackwell S, Beamon C, Szychowski JM, Andrews W; Cesarean Section Optimal Antibiotic Prophylaxis Trial Consortium. Risk Factors for Postcesarean Maternal Infection in a Trial of Extended-Spectrum Antibiotic Prophylaxis. Obstet Gynecol. 2017 Mar;129(3):481-485. doi: 10.1097/AOG.0000000000001899. PMID 28178058
- [Derived] Tita AT, Szychowski JM, Boggess K, Saade G, Longo S, Clark E, Esplin S, Cleary K, Wapner R, Letson K, Owens M, Abramovici A, Ambalavanan N, Cutter G, Andrews W; C/SOAP Trial Consortium. Adjunctive Azithromycin Prophylaxis for Cesarean Delivery. N Engl J Med. 2016 Sep 29;375(13):1231-41. doi: 10.1056/NEJMoa1602044. PMID 27682034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomly assigned to receive either azithromycin (at a dose of 500mg in 250 ml of saline, one time dose) or an identical-appearing saline placebo and the standard of care (cephazolin or clindamycin)
Pre-assignment Details: The addition of azithromycin and the standard of care (cephazolin or clindamycin) for antibiotic prophylaxis before cesarean delivery may further reduce the rate of postoperative infection. We evaluated the benefits and safety of azithromycin prophylaxis and the standard of care in women undergoing nonelective cesarean section.
Groups:
- Placebo and Standard of Care: Placebo: 250 cc normal saline Standard of care (cephazolin or clindamycin)
- Azithromycin and Standard of Care: Azithromycin: 500 mg in 250 cc normal saline 1 time dose and standard of care (cephazolin or clindamycin)
Period: Overall Study
Arm/Group | Placebo and Standard of Care | Azithromycin and Standard of Care
Started | 994 | 1019
Completed | 992 | 1018
Not Completed | 2 | 1
Not completed — Staff error, medication not administered | 1 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo With Standard Prophylaxis: Placebo: 250 cc normal saline Standard Prophylaxis: standard cephalosporin prophylaxis
- Azithromycin (Zithromax) With Standard Prophylaxis: Azithromycin: 500 mg in 250 cc normal saline 1 time dose Standard Prophylaxis: standard cephalosporin prophylaxis
- Total: Total of all reporting groups
Arm/Group | Placebo With Standard Prophylaxis | Azithromycin (Zithromax) With Standard Prophylaxis | Total
Number analyzed (Participants) | 994 | 1019 | 2013
Age, Continuous [Median (Standard Deviation); unit: years] | 28.4 (6.5) | 28.2 (6.1) | 28.3 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 994 | 1019 | 2013
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 994 | 1019 | 2013
Smoking Prevalence [Count of Participants; unit: Participants] | 122 | 97 | 219

OUTCOME MEASURES:

1. Primary Outcome: Participants With Endometritis and/or Wound Infection and/or Other Post-cesarean Infections (Occurring Within 6 Weeks of Delivery)
Description: Endometritis was defined as the presence of at least two of the following signs with no other recognized cause: fever (temperature of at least 38°C [100.4°F]), abdominal pain, uterine tenderness, or purulent drainage from the uterus. Wound infection was defined as the presence of either superficial or deep incisional surgical-site infection characterized by cellulitis or erythema and induration around the incision or purulent discharge from the incision site with or without fever and included necrotizing fasciitis. Wound hematoma, seroma, or breakdown alone in the absence of the preceding signs did not constitute infection.
Time Frame: Up to 6 weeks after delivery
Population: The specific characteristics related to the cesarean delivery, including indications for cesarean delivery, receipt of standard prophylaxis, timing of receipt of study medication, and type of surgical skin preparation, were similar in the two groups.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: 250 cc normal saline
  Placebo: 250 cc normal saline
- Azithromycin: Azithromycin: 500 mg in 250 cc normal saline 1 time dose
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 992 | 1018
Participants | 119 | 62

2. Other Pre Specified Outcome: Neonatal Morbidities (Listed Below)
Description: morbidities include: death, Respiratory Distress Syndrome (RDS), Bronchopulmonary Dysplasia (BPD), Periventricular Leukomalacia (PVL) suspected or proven sepsis, Necrotizing Enterocolitis (NEC) Intraventricular Hemorrhage (IVH) and systemic inflammatory response syndrome
Time Frame: Up to 3 months after birth
Measure: Count of Participants; unit: Participants
Groups:
- Placebo and Standard of Care: Placebo: 250 cc normal saline and standard of care (cefazolin or clindamycin)
- Azithromycin and Standard of Care: Azithromycin: 500 mg in 250 cc normal saline 1 time dose and Standard of Care (cefazolin or clindamycin
Arm/Group | Placebo and Standard of Care | Azithromycin and Standard of Care
Number analyzed (Participants) | 992 | 1018
Participants | 135 | 146

3. Other Pre Specified Outcome: Neonatal Intensive Care Unit (NICU) Admission
Description: Neonates who are admitted to the NICU due to morbidities diagnosed from birth and up to three months of life. Morbidities as defined in the Neonatal morbidities outcome measure.
Time Frame: Up to 3 months after birth
Measure: Count of Participants; unit: Participants
Groups:
- Azithromycin and Standard of Care: Azithromycin: 500 mg in 250 cc normal saline 1 time dose and Standard of care (cefazolin or clindamycin)
Arm/Group | Placebo and Standard of Care | Azithromycin and Standard of Care
Number analyzed (Participants) | 992 | 1018
Participants | 169 | 171

4. Other Pre Specified Outcome: Neonatal Readmission
Time Frame: Up to 3 months after birth
Population: Hospitalization after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo With Standard Prophylaxis | Azithromycin (Zithromax) With Standard Prophylaxis
Number analyzed (Participants) | 992 | 1018
Participants | 43 | 39

5. Other Pre Specified Outcome: Maternal Fever
Time Frame: Up to 6 weeks after delivery
Population: Postpartum Fever
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo With Standard Prophylaxis | Azithromycin (Zithromax) With Standard Prophylaxis
Number analyzed (Participants) | 992 | 1018
Participants | 81 | 51

6. Other Pre Specified Outcome: Maternal Postpartum Readmission or Unscheduled Visit
Description: Maternal postpartum unscheduled visit or readmission to the hospital
Time Frame: Up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Groups:
- Placebo and Standard of Care: Placebo: 250 cc normal saline Standard of care (cefazolin or clindamycin)
- Azithromycin and Standard of Care: Azithromycin: 500 mg in 250 cc normal saline 1 time dose Standard of care (cefazolin or clindamycin)
Arm/Group | Placebo and Standard of Care | Azithromycin and Standard of Care
Number analyzed (Participants) | 992 | 1018
Participants | 123 | 83

7. Other Pre Specified Outcome: Maternal Postpartum Antibiotic Use
Description: Maternal postpartum use of antibiotics
Time Frame: Up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo and Standard of Care | Azithromycin and Standard of Care
Number analyzed (Participants) | 992 | 1018
Participants | 166 | 126

8. Other Pre Specified Outcome: Maternal Serious Adverse Events
Description: All maternal serious adverse events
Time Frame: Up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo and Standard of Care | Azithromycin and Standard of Care
Number analyzed (Participants) | 992 | 1018
Participants | 29 | 15

9. Other Pre Specified Outcome: Neonatal Serious Adverse Events
Description: Composite for all neonatal serious adverse events
Time Frame: Up to 3 months after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo and Standard of Care | Azithromycin and Standard of Care
Number analyzed (Participants) | 992 | 1018
Participants | 5 | 7

10. Other Pre Specified Outcome: Infant Pyloric Stenosis
Description: Any diagnosis of pyloric stenosis based on clinical presentation and radiological and/or surgical confirmation
Time Frame: up to 3 months after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo and Standard of Care | Azithromycin and Standard of Care
Number analyzed (Participants) | 992 | 1018
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Up to 6 weeks after delivery
Description: Maternal serious adverse events (maternal safety composite outcome) included death, suspected allergic reactions (including anaphylaxis or generalized skin rash), any serious adverse event leading to the discontinuation of a study medication or suspected to be due to the medication, and any other reported serious adverse complication, including pulmonary embolism, admission to an intensive care unit (ICU), and cardiac events.
Groups:
- Azithromycin and Standard of Care: Azithromycin: 500 mg in 250 cc normal saline and Standard of care (cefazolin or clindamycin)
Arm/Group | Placebo and Standard of Care | Azithromycin and Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/992 | 0/1018
Serious Adverse Events (participants affected / at risk) | 29/992 | 15/1018
Other Adverse Events (participants affected / at risk) | 14/992 | 9/1018
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo and Standard of Care (N=992) | Azithromycin and Standard of Care (N=1018)
Severe allergic reaction (Immune system disorders) | 29 (29) | 15 (15) — Allergy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo and Standard of Care (N=992) | Azithromycin and Standard of Care (N=1018)
ICU admission (General disorders) | 14 (14) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No